CLINICAL TRIAL: NCT06033326
Title: Validation of the French Version of the Lithium Knowledge Test (LKT) for Patients Treated With Lithium in Psychiatric Unit Hospitals
Brief Title: Validation of the French Version of the Lithium Knowledge Test (LKT)
Acronym: LKT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_98
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Patient Treated With Lithium, With Bipolar or Schizo-affective Disorder, Hospitalized in a Psychiatric Ward
Keywords: Lithium; observance; security; Lithium Knowledge Test
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lithium is a drug used to treat several psychiatric illnesses. This medication requires particular vigilance because it has a narrow therapeutic margin: the dose necessary to obtain an effective treatment is close to the toxic dose.

The blood dosage of the drug and the patient's knowledge of the drug are necessary to optimize and secure the drug intake.

The objective of this observational study is to confirm that the score obtained by the LKT lithium knowledge self-questionnaire translated into French is representative of the knowledge of patients treated with lithium.

Participants will be asked to complete this questionnaire twice, and the scores obtained will be compared to the blood lithium level to see if a good score is associated with an effective blood lithium concentration.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in a psychiatric ward or in an EPSM for more than 10 consecutive days
* Patient treated with IR or ER lithium LI
* Patient over 18 years of
* Patient on a fixed dosage of lithium for more than 5 days prior to blood sampling for lithiaemia testing
* Obtain patient's non-opposition

Exclusion Criteria:

* Clinically unstable patient or patient with a cognitive disorder that makes it impossible to perform interview and/or completion of the LKT self-questionnaire
* Patients under guardianship or trusteeship
* Illiterate patients
* Patient with a therapeutic target concentration different from general recommendations (e.g. elderly subject)
* Patient receiving a pharmaceutical interview or any other interview between the completion of the 1 and 2nd questionnaires, likely to modify the LKT score.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in an adult psychiatric ward or staying in an EPSM in the cities included in this study
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of the factorial validity of the score from the first completed LKT self-questionnaire | 2 yaers
  Baseline: percentage of inertia explained by the first component of the principal component analysis Maximum time to obtain scores for 300 self-questionnaires: 2 years

SECONDARY OUTCOMES:
Evaluation of the internal consistency of the LKT score: is acceptable if Cronbach's alpha is greater than 0.7 | 2 yaers
  Baseline after data collection: percentage of inertia explained by the first component of the principal component analysis Maximum time to obtain scores for 300 self-questionnaires: 2 years
External validity of the LKT self-questionnaire by measuring the correlation between the lithiaemia assay at D0 and the score obtained on the self-questionnaire at D0. | 2 yaers
  Baseline after data collection: percentage of inertia explained by the first component of the principal component analysis Maximum time to obtain scores for 300 self-questionnaires: 2 years
Evaluation of the test/retest reliability of the LKT self-questionnaire score measured at D0 and D4. | 2 years
  Baseline and 4 days after data collection Maximum time to obtain scores for 300 self-questionnaires: 2 years
Comparison of lithiaemia at D0 between patients with good knowledge (i.e. a LKT self-questionnaire score at D0 > 6) and those with poor knowledge of treatment | 2 years
  Baseline and 4 days after data collection Maximum time to obtain scores for 300 self-questionnaires: 2 years
Search for factors associated with the LKT self-questionnaire score at J0. | 2 years
  Baseline and 4 days after data collection Maximum time to obtain scores for 300 self-questionnaires: 2 years